Title of the study: Partnership in Resilience for Medication Safety (PROMIS)

NCT number: <u>NCT05880368</u>

Date of approval by University of Texas Arlington Institutional Review Board (as IRB

Protocol #: 2019-0439.25): May 10, 2023



## The University of Texas at Arlington (UTA)

## **Verbal Consent Script for Post Visit Survey**

I am asking you to participate in a UT Arlington research study titled "Partnership in Resilience for Medication Safety." We are asking you to tell us about your visit experience today in a survey. This will take approximately 10 minutes. As compensation for your participation, you will be entitled to receive a \$10 Walmart gift card. This survey is part of a clinical trial. A description of this clinical trial will be available on http://www.ClinicalTrials.gov , as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

The survey is not expected to pose any risks beyond those that you would experience in your everyday life or during routine medical visits. The only potential risk to you would be a breach of confidentiality. However, the study investigators will take all precautions necessary to protect your confidentiality.

Your participation and answers will not affect the care you receive at this clinic. Your responses will not be shared with your provider or the clinic.

The decision to participate is entirely yours. If you feel uncomfortable answering some of the questions in the survey, you may skip them. You can also quit the survey at any time without any consequences.

Do you have any questions before proceeding to answering the survey?

You are indicating your voluntary agreement to participate in the PROMIS research project by beginning this survey.